CLINICAL TRIAL: NCT02372435
Title: Efficacy and Safety of Fast-track Treatment for Prosthetic Joint Infection (PJI)
Brief Title: Short Interval in Treatment of PJI
Acronym: Fast-track
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Andrej Trampuz, PD Dr. Andrej Trampuz, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ChariteU
Record Dates: First submitted 2015-01-23; First posted 2015-02-26 (Estimated); Last update posted 2015-02-26 (Estimated); Status verified 2015-02

CONDITIONS: Hip Prosthetic Joint Infection; Knee Prosthetic Joint Infection; Shoulder Prosthetic Joint Infection
Keywords: PJI

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Short interval (Experimental): Re-Implantation of the prosthesis after a short interval of 2-3 weeks after explantation ("fast-track-arm").
  Interventions: Procedure: Shortening of the interval of two-stage prosthesis exchange
- Long interval (Active Comparator): Re-Implantation of the prosthesis after a Long interval of 6-10 weeks (standard surgical treatment).
  Interventions: Procedure: Shortening of the interval of two-stage prosthesis exchange

INTERVENTIONS:
Procedure: Shortening of the interval of two-stage prosthesis exchange — The Intervention consist in shortening of the interval between Explantation and re-implantation in patients undergoing a two-stage prosthesis Exchange. Comparison between arms is performed between short and long interval before re-implantation.

SUMMARY:
Patients with hip, knee and shoulder PJI, will be treated with a two-stage exchange Revision.

Patients will be randomized into 2 groups: the experimental Group will get a reimplantation after a short interval (2-3 weeks) while the control Group after a long standard interval.

Primary objective of the study is "Infection outcome". The infection-free status is defined as absence of clinical (e.g. no fistula), laboratory (e.g. normal C-reactive protein) and radiological signs of infection (e.g. no septic loosening).

Secondary objective is "Functional outcome".The functional assessment will be performed using joint-specific scores (HARRIS HIP SCORE, CONSTANT SHOULDER SCORE, KNEE SOCIETY SCORE, OXFORD HIP SCORE, OXFORD KNEE SCORE, QUICK DASH SCORE) involving the range of motion (ROM), patient mobility / independency in daily life, subjective evaluation of pain using a visual analog pain scale (1-10 points) and life-quality evaluation (EQ5D5L score).

DETAILED DESCRIPTION:
A two-stage prosthesis exchange after a long interval of ≥6 weeks is considered the "gold standard" for management of prosthetic joint infection (PJI). We will compare the efficacy and safety of a novel surgical approach with short interval of 2-3 weeks ("fast-track") compared to the standard long interval of 6-10 weeks. Included will be patients with hip, knee or shoulder PJI, in whom all prosthetic components are removed; excluded will be patients treated with prosthesis retention or one-stage exchange and PJI caused by difficult-to-treat organisms. Patients will be randomized into short versus long interval surgical procedure, using a standard antibiotic regimen of 12 weeks in both study arms. The recruitment period of this multicenter treatment/outcome trial is 24 months, follow-up period 12 months and the calculated sample size 418 patients (i.e. 209 patient for each study arm). Primary endpoint is the infection outcome, secondary endpoint is the functional outcome, defined by established scores for joint-specific scores, pain and quality of life scores. The expected outcomes in the short interval ("fast-track") arm are (i) improved infection outcome (i.e. longer infection-free period and less treatment-related adverse events); (ii) improved functional outcome, and (iii) reduced healthcare expenses. In addition, pharmacokinetic studies will be performed and a biobank of microbes and biological samples will be established. This study has high clinical relevance for an increasing public health challenge related to device-associated infections.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged ≥18 years with hip, knee or shoulder PJI, in whom all prosthetic components are removed.
* The standard treatment for systemic and local antibiotics is followed (predetermined algorithm).
* Subjects are willing to participate in the study (signed informed consent) and comply with planned follow-up assessments (at 3, 6 and 12 months after study inclusion).

Exclusion Criteria:

* Treatment with debridement and prosthesis retention (e.g. performed in early postoperative or acute hematogenous infections with symptom duration <3 weeks) or one-stage exchange.
* PJI caused by difficult-to-treat organisms, including rifampin-resistant staphylococci, quinolone-resistant Gram-negative bacilli and fungi.
* Subject previously enrolled in this study or is currently enrolled in another competitive investigational study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 418 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Infection outcome | 12 months after surgery
  Duration of infection-free interval and frequency of adverse events related to surgical treatment. The infection-free status is defined as absence of clinical (e.g. no fistula), laboratory (e.g. normal C-reactive protein) and radiological signs of infection (e.g. no septic loosening).

SECONDARY OUTCOMES:
Functional outcome | 12 months after surgery
  The functional assessment will be performed using joint-specific scores (HARRIS HIP SCORE, CONSTANT SHOULDER SCORE, KNEE SOCIETY SCORE, OXFORD HIP SCORE, OXFORD KNEE SCORE, QUICK DASH SCORE) involving the range of motion (ROM), patient mobility / independency in daily life, subjective evaluation of pain using a visual analog pain scale (1-10 points) and life-quality evaluation (EQ5D5L score).

CONTACTS AND LOCATIONS:
Overall Officials: Andrej Trampuz, PD, Principal Investigator — Charite University, Berlin, Germany